CLINICAL TRIAL: NCT03705663
Title: Identification of the Pre-exposure Prophylaxis (PrEP) Cascade for Women and Integration of PrEP Into Women's Family Planning Services: a Prospective Cohort
Brief Title: Identification of the Pre-exposure Prophylaxis (PrEP) Cascade for Women.
Acronym: PrEP
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0870
Record Dates: First submitted 2018-09-21; First posted 2018-10-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Pre-Exposure Prophylaxis
Keywords: HIV prevention, PrEP cascade, women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dried Blood Spots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women interested in HIV PrEP: Cis-gender women at high risk for HIV interested in or initiating HIV PrEP
  Interventions: Behavioral: PrEP initiation

INTERVENTIONS:
Behavioral: PrEP initiation — Women who are interested in or who initiate PrEP will be followed in a prospective cohort to identify and populate the PrEP cascade for cis-gender, high risk women

SUMMARY:
Pre-exposure prophylaxis (PrEP) is a daily pill that greatly reduces the risk of transmission of human immunodeficiency virus (HIV), however the barriers to PrEP use for women are understudied and PrEP is underutilized by women. Partnering with the DC Department of Health and the DC Center for AIDS Research (DC-CFAR), the overarching goals are (1) to identify and populate the PrEP cascade for women, (2) to provide a blueprint for family planning providers to integrate HIV prevention into their practices and target evidence-based interventions to the women at highest risk for HIV in their communities, and (3) to evaluate the cost-effectiveness of this intervention. The overarching hypotheses are that (1) the timeline and roadmap to PrEP adoption and the PrEP cascade will be different for cis-gender women than that described for men who have sex with men (MSM) and transgender women, (2) women seeking family planning services will be eligible for and interested in PrEP and family planning providers are ideally situated to provide this care, and (3) provision of PrEP in the family planning setting will be cost-effective. This research proposes to evaluate (1) PrEP cascade of events for women (eligibility for PrEP, acceptability/interest in PrEP, access/linkage to a PrEP program, initiation of PrEP, retention, and adherence to PrEP) and (2) the integration of universal screening for PrEP and PrEP provision into a women's family planning clinic. This research will allow for targeted evidence-based interventions to reach women at high-risk for HIV and will provide a blueprint for the implementation of PrEP services in the family planning setting nationally.

DETAILED DESCRIPTION:
Pre-exposure prophylaxis (PrEP) with daily tenofovir-emtricitabine (TFV/FTC) reduces transmission of human immunodeficiency virus (HIV) by up to 92%, however PrEP is underutilized, especially in women. Women account for nearly 20% of new HIV diagnoses-- most via heterosexual transmission; African-American women and women of color are disproportionately affected. PrEP is recommended for all women who "engage in sexual activity in a high prevalence area" and inconsistently use condoms. Despite this recommendation and local and national efforts to curb the HIV epidemic in the United States (US), PrEP has not been widely offered to high-risk cis-gender women and their "PrEP cascade" of events (eligibility for PrEP, acceptability/interest in PrEP, access/linkage to a PrEP program, initiation of PrEP, retention, and adherence to PrEP) for women has not been described in order to inform intervention.

PrEP is especially critical for high-risk women in Washington DC (DC), an epicenter of the HIV epidemic in the US. Recent focus groups with African-American women at risk for HIV in DC revealed inadequate knowledge about and difficulty accessing PrEP, but high levels of acceptability and interest. Qualitative research and the research team's clinical initial experience in PrEP provision demonstrate that cis-gender women require more contact with providers and have more concerns regarding logistics, interactions, and disclosure of PrEP use to partners compared to transgender women and men who have sex with men (MSM)-suggesting 1) a different timeline for initiation of PrEP and 2) a different PrEP cascade in women. Identifying and populating the PrEP cascade for women will allow the investigators to target evidence-based interventions to reach women at risk for HIV.

The same high-risk sexual activity that puts women at risk for HIV also puts women at risk for unintended pregnancy; the latter leads many of them to seek care in family planning clinics. While there may be synergies in offering PrEP along with contraception and pregnancy termination services at family planning clinics, most family planning clinics do not offer PrEP. A recent study demonstrated low levels of PrEP knowledge and of comfort prescribing PrEP among family planning providers, however 90% of providers reported interest in learning more about PrEP and the majority of family planning patients surveyed reported they would consider using PrEP. The investigators hypothesize that integrating HIV prevention into family planning services would empower women and better meet their preventative health needs.

Partnering with the DC Department of Health (DOH) and the DC Center for AIDS Research (DC-CFAR), the over-arching goals are (1) to identify and populate the PrEP cascade for women, (2) to provide a blueprint for family planning providers to integrate HIV prevention into their practices and target evidence-based interventions to the women at highest risk for HIV in their communities, and (3) to evaluate the cost-effectiveness of this intervention. The overarching hypotheses are that (1) the timeline and roadmap to PrEP adoption and the PrEP cascade will be different for cis-gender women than that described for MSM and transgender women, (2) women seeking family planning services will be eligible for and interested in PrEP and family planning providers are ideally situated to provide this care, and (3) provision of PrEP in the family planning setting will be cost-effective. MedStar Washington Hospital Center (MWHC) provides the ideal setting to elucidate the PrEP cascade in women and to design and evaluate integrated PrEP services in the family planning setting. The Family Planning and Preventative Care (FPPC) clinic at MWHC provides over 800 family planning visits annually, the majority to African-American, low socioeconomic status women at high-risk for HIV. Family planning providers at MWHC are not yet routinely assessing PrEP eligibility or prescribing PrEP, however, the investigators anticipate that the majority of patients seeking care at FPPC will be eligible for and could benefit from PrEP. The investigators propose a prospective cohort to evaluate the following specific aims:

Specific Aim 1 To test the hypothesis that the PrEP cascade for women will be different than that described for men, the investigators will identify and populate the PrEP cascade by assessing women's risk factors for and perceived vulnerability to HIV, PrEP acceptability, initiation, continuation, and adherence. The investigators will describe the timeline and roadmap to PrEP uptake and will explore determinants of the stages of the PrEP cascade.

Specific Aim 2 To test the hypotheses that (a) family planning clinics provide a high-yield and feasible venue in which to reach women at high-risk for HIV acquisition and to offer PrEP initiation and follow-up, and (b) provision of PrEP in the family planning setting will be cost-effective, the investigators will assess the reach, effectiveness, adoption, implementation, maintenance (RE-AIM)[8], and cost-effectiveness of the integration and provision PrEP in a family planning clinic.

These results will overcome the primary obstacle to more effective provision of PrEP to high-risk cis-gender women by describing the PrEP cascade, which is needed to inform HIV prevention for women. Additionally, this study will provide critical insight into the provision of PrEP in a novel and practical setting. These results will lead directly to evidence based PrEP programs that can be integrated into family planning care nationally in high-risk areas, thereby addressing persisting disparities in gender and race in HIV prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Cis-gender women
2. Interested in PrEP and/or initiating PrEP

Exclusion Criteria:

1. HIV positive
2. Severe liver disease
3. Severe renal (kidney) disease
4. Signs/symptoms of acute HIV infection (such as fever, swollen lymph nodes, sore throat, skin rash, body aches)
5. Do not speak English or Spanish
6. No access to a telephone for follow-up
7. Planning to leave the Washington, DC area in the next 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender women
Study Population: Women at high risk for HIV interested in and/or initiating pre-exposure prophylaxis (PrEP)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
PrEP cascade in cis-gender women | 2 years
  We will be using a variety of measures to describe the "PrEP cascade" for women, specifically the proportion of women who initiate, continue, and adhere to PrEP and the timeline associated with the steps of the PrEP cascade.

SECONDARY OUTCOMES:
Implementation analysis of universal PrEP screening | 2 years
  Descriptive implementation analysis using the RE-AIM framework:
  Reach - The absolute number/proportion/representativeness of women who initiate PrEP, continue PrEP etc.
  Efficacy - The impact of universal PrEP screening on PrEP initiation and HIV prevention.
  Adoption - The absolute number/proportion/representativeness of clinics/providers who are willing to initiate universal PrEP Implementation - At the setting level, the providers' fidelity to the intervention's protocol. At the individual level, implementation refers to women's PrEP uptake.
  Maintenance - The extent to which the PrEP program becomes institutionalized or part of the routine organizational practices and policies. Within the RE-AIM framework, maintenance also applies at the individual level, defined as the long-term effects of a program on outcomes after 6 or more months after the most recent intervention contact-in this case continuation of PrEP
Cost effectiveness analysis of universal PrEP screening | 2 years
  Cost-effectiveness analysis of the integration and provision PrEP in a family planning clinic using quality adjusted life years (QALY) and cost.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel K Scott, MD, Principal Investigator — Medstar Health Research Institute
Locations (2):
- United States (2):
  - DC Health and Wellness Center, Washington D.C., District of Columbia
  - Rachel Scott, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Yes
Sharing of our data on 1) the PrEP cascade for women and 2) the integration of PrEP provision into the family planning setting that will result from this proposed study is an integral part of both our proposed research activities and planned next steps. We plan to make our results available both to the community of clinicians and researchers interested in HIV prevention in women and/or the integration of PrEP in the family planning setting to avoid duplication of research, to allow the clinical and research community to benefit from the novel conclusions and insights that may arise from this research, and to foster research collaboration with other sites to build upon our findings.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon request.
Access Criteria: Pending review of concept sheet.

REFERENCES:
- [Derived] Scott RK, Deyarmond M, Marwitz S, Huang JC, Moriarty P, Visconti AJ, Beverley J, Elion R, Coleman M, Hull SJ. Implementation of an Educational Intervention to Improve HIV Pre-Exposure Prophylaxis Services for Women in an Urban Sexual Health Clinic. AIDS Patient Care STDS. 2023 Sep;37(9):447-457. doi: 10.1089/apc.2023.0107. PMID 37713289